CLINICAL TRIAL: NCT06185283
Title: Milled in Versus Round Bar for Mini-implant Retained Mandibular Overdentures :A8 Year Retrospective Study of Peri-implant Bone Changes and Posterior Ridge Resorption
Brief Title: Milled in Versus Round Bar for Mini-implant Retained Mandibular Overdentures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: M01010023RP
Record Dates: First submitted 2023-12-03; First posted 2023-12-29 (Actual); Last update posted 2023-12-29 (Actual); Status verified 2023-11

CONDITIONS: Bone Loss
Keywords: milled bar; round bar
MeSH Terms: conditions — Bone Diseases, Metabolic

STUDY DESIGN:
Intervention Model Description: A convenience sample of 18 completely edentulous participants were selected for this retrospective study from patients originally available at the start of the trial .
  The patients were equally divided into two groups at the start of the trial. The patients (average age 45-60 years) were selected for this study from outpatient clinic of Removable Prosthodontics Department, Faculty of Dentistry, Mansoura University
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- milled bar group (Other): . O-Ball impression copings were snapped directly onto each O-Ball mini dental Implants. A Pick-Up closed tray impression technique was made using polyether impression material. MDI Lab Analog was pressed into the coping until a snap fit was observed .The impression was poured into dental stone to form a stone model for scanning
  The cast was scanned using 3SHAPE TRIOS and the bar constructed throughout the production steps:
  Step 1: Order Creation ,Step 2: scan the lab analog of MDI on the stone model scanned with D700 scanner. Step 3: CAD Designing (first select preparation in teeth view from canine to canine-click abutment button-choose restoration type (bar)-choose restoration material (wax) .Step 4: Sending to CAM for Manufacturing, Step 5: Manufacturing (cutting from disc of modeling wax).
  Interventions: Diagnostic Test: panoramic x-ray
- round bar (Other): Prefabricated plastic bar pattern (RHIN 83 OT BAR multi use) was pre scanned for standardization of all cases. After cast scanning the abutment copy was designed and again standardized for all MDI. The pre scanned bar was inserted over the copies. The same procedure for manufacturing was followed as that of milled -in bar.
  The finished bar is brought to the patient's mouth, seated accurately. The denture is then tried, fitted and extensions adjusted in the usual manner. The denture fitting surface was; the hygienic space under the bar was blocked-out with wax.
  plastic clip was adapted to their metal sleeve, adapted to the bar, the occlusion was checked and then they were picked-up using auto-polymerized acrylic resin while the patient was instructed to close lightly in centric occlusion. After finishing and polishing procedures, the mandibular denture was clinically remounted to adjust any interferences in the centric and eccentric the occlusal contacts.
  Interventions: Diagnostic Test: panoramic x-ray

INTERVENTIONS:
Diagnostic Test: panoramic x-ray — Long cone paralleling technique and a film holder designed specifically for implant imaging were used for intraoral radiograph. To maintain the same film- implant distance and cone implant distance, a modification were carried out for the film holder. This modification is a hole drilled exactly above the implant fixture so the distance were maintained during subsequent film exposures. Through this modification, standardized radiographs were achieved.
  Other Names: periapical x-ray

SUMMARY:
purpose: The primary purpose of this retrospective radiographic study were conducted to compare between milled bar and round bar for mini implant retained overdentures (IODs) on peri-implant bone changes and posterior mandibular ridge resorption .Study Design: A convenience sample of 18 completely edentulous participants were selected for this retrospective study from patients originally available at the start of the trial .

The null hypothesis was that there were no significant difference between milled in and round bar attachment retained implant supported overdentures in posterior ridge resorption and peri-implant bone changes.

DETAILED DESCRIPTION:
Study Design:

A convenience sample of 18 completely edentulous participants were selected for this retrospective study from patients originally available at the start of the trial. The patients were informed about the study objectives and they were signed an informed consent and the protocol were approved by the Ethical Committee, Faculty of Dentistry, Mansoura University.

The patients were equally divided into two groups at the start of the trial. The patients (average age 45-60 years) were selected for this study from outpatient clinic of Removable Prosthodontics Department, Faculty of Dentistry, Mansoura University.

Patients' criteria:

Completely edentulous maxillary and mandibular residual alveolar ridges covered with healthy mucosa without any remaining roots or local inflammation as detected by digital panoramic x-ray and clinical examination.. Anterior mandibular bone length was sufficient to allow proper implant placement as assessed by digital panoramic radiograph. Patients were of class I Angel's maxillo-mandibular relation with at least 22mm of restorative space allow for bar construction as detected by tentative jaw relation, and good bone quality (classes 1 to 3 according to Lekholm and Zarb). Participants with diabetes mellitus, osteoporosis, immunological dysfunction, anticoagulant medication, radiation to the head and neck region, smoking habits ,and systemic diseases that interfere with implants osseointegration were excluded from the study .For each patient, overdentures assisted by four splinted mini dental implants According to type of bar attachment used for splinting the four MDIs, patients were divided into two equal groups where: Group I: Received milled-in bar and Group II: Received round bar joint attachment. O-Ball impression copings were snapped directly onto each O-Ball MDI Implant. A Pick-Up closed tray impression technique was made using polyether impression material. MDI Lab Analog was pressed into the coping until a snap fit was observed .The impression was poured into dental stone to form a stone model for scanning Bar construction

Milled-in bar construction for group I:

The cast was scanned using 3SHAPE TRIOS and the bar constructed throughout the production steps:

Step 1: Order Creation ,Step 2: scan the lab analog of MDI on the stone model scanned with D700 scanner. Step 3: CAD Designing (first select preparation in teeth view from canine to canine-click abutment button-choose restoration type (bar)-choose restoration material (wax) .Step 4: Sending to CAM for Manufacturing, Step 5: Manufacturing (cutting from disc of modeling wax). After casting into cobalt chromium alloy, the metal bar was secured into position on the cast and adjusted to the table of the milling machine. The facial and lingual guide planes were refined and the bar was finished and polished to a high shine.

Round bar fabrication for group II:

Prefabricated plastic bar pattern (RHIN 83 OT BAR multi use) was pre scanned for standardization of all cases. After cast scanning the abutment copy was designed and again standardized for all MDI. The pre scanned bar was inserted over the copies. The same procedure for manufacturing was followed as that of milled -in bar.

The finished bar is brought to the patient's mouth, seated accurately. The denture is then tried, fitted and extensions adjusted in the usual manner. The denture fitting surface was; the hygienic space under the bar was blocked-out with wax.

For group I: Metallic Retentive clips were directly fastened to the bar. After the occlusion was rechecked, the clips were picked-up using auto-polymerized acrylic resin while the patient was instructed to close lightly in centric occlusion.

For group II: plastic clip was adapted to their metal sleeve, adapted to the bar, the occlusion was checked and then they were picked-up using auto-polymerized acrylic resin while the patient was instructed to close lightly in centric occlusion. After finishing and polishing procedures, the mandibular denture was clinically remounted to adjust any interferences in the centric and eccentric the occlusal contacts.

The prosthodontic maintenance required for the IODs and opposing dentures were evaluated during a 8-year follow-up period and compared between the 2 bar design attachments for IODs.

Patients' evaluation

Radiographic Evaluation of peri-implani bone changes:

A. Long cone paralleling technique and a film holder designed specifically for implant imaging will be used for intraoral radiograph. To maintain the same film- implant distance and cone implant distance, a modification will be carried out for the film holder. This modification is a hole drilled exactly above the implant fixture so the distance will be maintained during subsequent film exposures. Through this modification, standardized radiographs will be achieved.

B. The long cone periapical radiographs will be taken using a digital photostimulable phosphor plate (PSP) aligned parallel to the implant and all radiographs will be taken by the same standard intraoral X-ray machine with exposure settings of 60 kV, 7 mA for 0.16 s. Subsequently, lines and reference points will be marked. Detect magnification error by comparing the implant dimensions in the radiographs with the actual implant dimensions this ratio allow us to obtain the actual values of the bone changes.

C. For marginal alveolar bone changes, the distance between implant shoulder (A) and first bone to implant contact (B) indicated vertical bone level (DIB) in mm. Vertical bone loss (VBL) will be calculated by subtracting DIB at (T8) from DIB at T0. Alveolar bone changes will be measured mesially and distally. B. periapical x-ray will be done immediately at insertion (T0) ,the second one (T3), and after 8 years following the insertion (T8).

Evaluation of Posterior Mandibular Alveolar Bone Changes:

Posterior area index will be evaluated by proportional measurement of a posterior mandibular area like the method described by Wright and Watson. Two panoramic radiographs will be taken, one at time of insertion (T0) and the second one after 8 years following the insertion (T8). The reference points and lines will traced using AutoCAD 2018 software.

The posterior mandibular area will outline by joining points at the gonion (G/G') to the lower border of the mental foramen (M/M') and the sigmoid notch (S/S'). (N/N') representing the center of the triangle joining the three points M-S-G/M'-S'-G'. Reference area will be represented by a line joining M-G-N/M'-G'-N'. The experimental area will determined A-P-G-M/A'-P'-G'-M' where A-L/A'-L' represents the crest of the mandibular ridge to the lower border of the mandible and perpendicular to the M-G/M'G' line. The area difference which represents the bone resorption will be calculated by the equation (X/Y+X'/Y')/2 where X/X' represents the experimental area and Y/Y' represents the reference area.

ELIGIBILITY:
Inclusion Criteria:

* Completely edentulous maxillary and mandibular residual alveolar ridges covered with healthy mucosa without any remaining roots or local inflammation as detected by digital panoramic x-ray and clinical examination.. Anterior mandibular bone length was sufficient to allow proper implant placement as assessed by digital panoramic radiograph. Patients were of class I Angel's maxillo-mandibular relation with at least 22mm of restorative space allow for bar construction as detected by tentative jaw relation, and good bone quality (classes 1 to 3 according to Lekholm and Zarb).

Exclusion Criteria:

* Participants with diabetes mellitus, osteoporosis, immunological dysfunction, anticoagulant medication, radiation to the head and neck region, smoking habits ,and systemic diseases that interfere with implants osseointegration were excluded from the study

Ages: 45 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2020-04-11 (Actual); Study Completion 2023-09 (Actual)

PRIMARY OUTCOMES:
peri-implant bone loss | 8 year
  For marginal alveolar bone changes, the distance between implant shoulder (A) and first bone to implant contact (B) indicated vertical bone level (DIB) in mm. Vertical bone loss (VBL) were calculated by subtracting DIB at (T8) from DIB at T0. Alveolar bone changes were measured mesially and distally. B. periapical x-ray were done immediately at insertion (T0) ,the second one (T3) Two panoramic radiographs were taken, one at time of insertion (T0) and the second one after 8 years following the insertion (T8). The reference points and lines were traced using AutoCAD 2018 software
posterior ridge resorption | 8 year
  for posterior area in mandible

CONTACTS AND LOCATIONS:
Overall Officials: Nermeen E Elkhamisy, Phd, Study Chair — Mansoura University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fromentin O, Lassauzay C, Abi Nader S, Feine J, de Albuquerque Junior RF. Testing the retention of attachments for implant overdentures - validation of an original force measurement system. J Oral Rehabil. 2010 Jan;37(1):54-62. doi: 10.1111/j.1365-2842.2009.02020.x. Epub 2009 Nov 11. PMID 19912482
- [Derived] El-Khamisy NES, Emera RMK, Awad HN. Milled in versus round bar for mini implant retained mandibular overdentures: a 8-year retrospective radiographic study of peri-implant bone changes and posterior ridge resorption. BMC Oral Health. 2025 Aug 16;25(1):1334. doi: 10.1186/s12903-025-06689-6. PMID 40818957